CLINICAL TRIAL: NCT02825550
Title: Radiopaque Microsphere (Hydrophilic Series) for Hepatoma Embolization Therapy
Brief Title: Taiwan ACE Beads for Hepatoma Embolization Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Collaborators: The Industrial Technology Research Institute (Other); National Cheng Kung University (Other); National Research Program for Biopharmaceuticals, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-104-046
Record Dates: First submitted 2016-06-02; First posted 2016-07-07 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Cancer of Liver
Keywords: Hepatoma; Transcatheter Arterial chemo-embolization; Microsphere
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hepatoma treated using Taiwan ACE Beads (Experimental): The use of Taiwan ACE Beads (T-ACE) microspheres embolization as a treatment for patients with hepatoma.
  Interventions: Device: Taiwan ACE Beads

INTERVENTIONS:
Device: Taiwan ACE Beads — Similar with conventional TACE, radiologist inject lipiodol with doxorubicin first, then use Taiwan ACE Beads instead of Gelfoam or polyvinyl alcohol.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Radiopaque Microsphere (T-ACE Beads) interventional therapy for patients with liver cancer

DETAILED DESCRIPTION:
The study will evaluate the safety and tolerability of Taiwan ACE Beads used for chemoembolization for the treatment of unresectable hepatocellular carcinoma.

The investigators will study the overall response rates of lesions with Taiwan ACE Beads. The procedure is similar with conventional TACE (transcatheter arterial chemoembolization). At the target vessels, radiologists will inject lipiodol with doxorubicin first, then Taiwan ACE Beads instead of Gelfoam or PVA (polyvinyl alcohol). The end point of injection is also similar with conventional TACE.

Determine the complication rates, progression free survival (PFS) and overall survival (OS) following Taiwan ACE Beads embolization.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria in order to be entered into the study:

A. Both genders of patients age 18 or older.

B. Patients diagnosed of liver cancer (MUST meet at least ONE of the following criteria:)

1. Diagnosed via tumor biopsy by Pathologists, and confirmed by on-service physician.
2. High risk patients (Viral hepatitis B or C or cirrhotics) with typical liver cancer image appeared on more than two radiographic examinations (Ultrasound, MRI, CT scan or Angiography).
3. High risk patients (Viral hepatitis B or C cirrhotics) with evidence of enlarging image of liver cancer via more than two follow-up records.

C. In intermediate stage by BCLC staging, tumor size between 3 to 6 centimeters, with liver function at Child-Pugh class<9, and is either difficult to accept an operation or reluctant to accept any operation.

D. Disease can be treated by transarterial chemoembolization, and can be evaluated by Ultrasound, Magnetic resonance imaging (MRI), or computed tomography (CT).

E. Performance status ECOG 2 or less. Patient has a life expectancy of at least 3 months.

Exclusion Criteria:

If patients meet any of the following criteria they may not be entered into the study:

A. major branch of portal vein has been invaded already; extrahepatic metastasis or the the other malignant tumors.

B. Evidences of decompensation: Total Bilirubin>2, PT prolong>3 seconds, AST > 500U/L, ALT> 500U/L, Child-Pugh class≧9, refractory ascites, active bleeding, hepatic encephalopathy, and severe infection.

C. Tumor size (diameter) larger than 6 centimeters or smaller than 3 centimeters.

D. Cr>2.0 mg/dL and eGFR<50%.

E. Allergic to iodine or other injections.

F. Other main organ failure (Heart, Lung, or Kidney)

G. WBC<3000, ANC<1500.

H. Performance status ECOG of 3 or more.

I. Unable to follow-up by ultrasound or CT scan.

J. Unwilling to sign a written informed consent form.

K. Pregnant women and breath feeding women.

L. Patients whose blood vessel are too difficult to do Taiwan ACE Beads procedure.

M. Prominent AV shunt.

N. Severe atherosclerosis.

O. Vasospasm or possible major vascular injury.

P. Arteriovenous shunt patients, diameter larger than the size of microsphere available.

Q. Collateral vascular exists and may endanger non-targeted area during arterial chemoembolization.

R. Contraindications for doxorubicin.

S. Number of tumors more than 3 and locate at different lobes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xi-Zhang Lin, Study Director — Department of Internal Medicine, National Cheng Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu YS, Lin XZ, Tsai HM, Tsai HW, Chen GC, Chen SF, Kang JW, Chou CM, Chen CY. Development of biodegradable radiopaque microsphere for arterial embolization-a pig study. World J Radiol. 2015 Aug 28;7(8):212-9. doi: 10.4329/wjr.v7.i8.212. PMID 26339465
- [Background] Chen CY, Liu HS, Lin XZ. Hydrodynamics-based gene delivery to the liver by bile duct injection of plasmid DNA--the impact of lasting biliary obstruction and injection volume. Hepatogastroenterology. 2005 Jan-Feb;52(61):25-8. PMID 15782986
- [Background] Luo TY, Shih YH, Chen CY, Tang IC, Wu YL, Kung HC, Lin WJ, Lin XZ. Evaluating the potential of (188)Re-ECD/lipiodol as a therapeutic radiopharmaceutical by intratumoral injection for hepatoma treatment. Cancer Biother Radiopharm. 2009 Oct;24(5):535-41. doi: 10.1089/cbr.2008.0603. PMID 19877883

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment started in April, 2016. The location was all taken place in National Cheng Kung University Hospital. Patients who met inclusion criteria were recruited.
Groups:
- Hepatoma Patients Treated With T-ACE Beads: In the Hepatoma Embolization Therapy, the catheter was placed to the appropriate position in tumor-supplying artery. Lipiodol containing doxorubicin were firstly injected, followed by the injection of our T-ACE beads-H series microspheres. The follow-up blood tests and adverse events were conducted afterwards. CT scan or MRI would be scheduled at the first and the third months to evaluate the change of tumor size.
Period: Overall Study
Arm/Group | Hepatoma Patients Treated With T-ACE Beads
Started | 13
Completed | 12
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Hepatoma Treated Using Taiwan ACE Beads: Clinical information of T-ACE beads H-series: Gender Male/Female 7/5, Age 71±8. The initial number of participants in the study was 13. However, one patient's blood test did not meet the standard before the operation, which led to his/her withdrawal from the clinical trial. Consequently, the total number of participants analyzed was 12.
Arm/Group | Hepatoma Treated Using Taiwan ACE Beads
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Region of Enrollment [Number; unit: participants]
  Taiwan | 12

OUTCOME MEASURES:

1. Primary Outcome: Patients Survival (Safety)
Description: Survival rate was evaluated since treatment day until the date of death or final observation.
Time Frame: An average of 12 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Hepatoma Treated Using Taiwan ACE Beads: Hepatoma patients received Taiwan ACE Beads (T-ACE) microspheres embolization to treat the tumors.
  Taiwan ACE Beads: The procedure is similar with conventional TACE. Radiologist inject lipiodol with doxorubicin first, then use Taiwan ACE Beads instead of Gelfoam or polyvinyl alcohol.
  Survival rate was evaluated since beginning of treatment until date of death or final observation.
Arm/Group | Hepatoma Treated Using Taiwan ACE Beads
Number analyzed (Participants) | 12
Participants | 12

2. Primary Outcome: Tumor Response (Efficacy)
Description: mRECIST criteria was used to evaluate tumor response in patients with hepatoma who received Taiwan ACE beads (T-ACE) microspheres embolization.
Time Frame: Before treatment, one month and three month after T-ACE using CT scan and MRI
Measure: Count of Participants; unit: Participants
Groups:
- Hepatoma Patients Treated With T-ACE Beads: We have 7 male and 5 female patients eligible in this study, HBV 4+1, HCV5+1, non-HBV and non-HCV 2, mean age 71± 8. Two patient received treatment at the first time. The other 10 patients received RFA 13 times, and TACE 23 times, and surgery 2 times. The response of the target lesions are: CR 3 PR 4 SD 3 PD 2 (for target lesions), and CR 2 PR 3 SD 3 PD 4 (for the overall response). Liver function, serological ALT(35±24) had mild elevation on the second day (61±47), but all return to baseline (40±20). AFP decreased from 168± 382 to 156± 264. [Conclusion] Our T-ACE Beads are safe and has some effects in treating hepatoma patients.For further clinical trials, loading appropriate chemotherapeutic agents to our microspheres for TACE is needed.
Arm/Group | Hepatoma Patients Treated With T-ACE Beads
Number analyzed (Participants) | 12
Participants
  Target Lesions: Complete Remission (CR) | 3
  Target Lesions: Partial Response (PR) | 4
  Target Lesions: Stable Disease (SD) | 3
  Target Lesions: Progressive Disease (PD) | 2
  Overall Response: Complete Remission (CR) | 2
  Overall Response: Partial Response (PR) | 3
  Overall Response: Stable Disease (SD) | 3
  Overall Response: Progressive Disease (PD) | 4

3. Secondary Outcome: Serum Level of AFP
Description: Serum Level of AFP [Time Frame: Baseline serum AFP levels (168±383) compared with one or three months of serum levels of AFP (144±256) after Taiwan ACE Beads procedure]
Time Frame: Baseline serum AFP levels compared with one or three months of serum levels of AFP after Taiwan ACE Beads procedure
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Hepatoma Treated Using Taiwan ACE Beads: Hepatoma patients received Taiwan ACE Beads (T-ACE) microspheres embolization to treat the tumors.
  Taiwan ACE Beads: The procedure is similar with conventional TACE. Radiologist inject lipiodol with doxorubicin first, then use Taiwan ACE Beads instead of Gelfoam or polyvinyl alcohol.
Arm/Group | Hepatoma Treated Using Taiwan ACE Beads
Number analyzed (Participants) | 12
ng/mL
  Baseline serum AFP levels | 168 (383)
  one or three months of serum levels of AFP | 144 (256)

ADVERSE EVENTS:
Groups:
- Adverse Event: There was no adverse event reported in this trial.
Arm/Group | Adverse Event
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
1. Case number : only 12 patients completed trial.
2. Tumor size limited to 3-6 cm only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No